CLINICAL TRIAL: NCT05511740
Title: Influence of Radiation Patterns Following Circadian Rhythm Upon Response of Radiotherapy of Uterine Cervical Cancer : Melatonin as a Radiosensitivity and Biological Marker
Brief Title: Circadian as A Prognostic Factor For Radiation Response in Cervical Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Irwan Ramli, Sp.Onk. Rad(K), Consultant of Radiation Oncology, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 27/PT02.FK/ETIK/2010
Record Dates: First submitted 2022-08-11; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Cervical Cancer; Radiotherapy Side Effect
Keywords: Radiosensitivity; Circadian rhythm
MeSH Terms: conditions — Uterine Cervical Neoplasms; Radiation Injuries

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning Radiation (No Intervention)
- Afternoon Radiation (Active Comparator)
  Interventions: Radiation: Afternoon Radiation

INTERVENTIONS:
Radiation: Afternoon Radiation — Melatonin, a hormone of the pineal gland, which levels are characteristic of circadian patterns, regulated with low levels of excretion in the afternoon, rises gradually during the night, peaks at dawn, and falls back in the afternoon and late afternoon. Many studies prove the function and potential of melatonin as circadian biomarkers and well correlated with the development of cancer.The function of melatonin is as an antiproliferation substance or hormone, induces apoptosis, inhibits invasion and metastasis.
  Arms: Afternoon Radiation

SUMMARY:
The study was a Randomized Clinical Trial (RCT) or clinical trial comparing the results of radiation treatment of 2 treatment groups, i.e. subject groups irradiated in the morning and in the afternoon, to check melatonin levels in cervical cancer patients. Since it is known that the function of melatonin is as an antiproliferation substance or hormone, induces apoptosis, inhibits invasion and metastasis.

ELIGIBILITY:
Inclusion Criteria:

* cervical cancer patients stage IIB-IIIB (FIGO)
* no previous treatment
* histopathologic examination results of squamous cell carcinoma (SCC)
* KPS > 70 with levels of Hb > 10 g%,

Exclusion Criteria:

* Distant metastasis and locally spread to the adjacent healthy tissue (urinary bladder or rectum).

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Radiation response | Four weeks after the completion of radiation
  We assessed the change in tumor size between the initial examination and the fourth week after the completion of irradiation, to classify the tumor response based on the modified WHO criteria which categorized as good response or poor response.

CONTACTS AND LOCATIONS:
Overall Officials: Irwan Ramli, MD, Principal Investigator — Department of Radiation Oncology Cipto Mangunkusumo Hospital

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: starting 6 months after publication
Access Criteria: requested via email

REFERENCES:
- [Result] Jung B, Ahmad N. Melatonin in cancer management: progress and promise. Cancer Res. 2006 Oct 15;66(20):9789-93. doi: 10.1158/0008-5472.CAN-06-1776. PMID 17047036
- [Result] Karbownik M, Reiter RJ. Melatonin protects against oxidative stress caused by delta-aminolevulinic acid: implications for cancer reduction. Cancer Invest. 2002;20(2):276-86. doi: 10.1081/cnv-120001154. PMID 11901547
- [Result] Vijayalaxmi, Thomas CR Jr, Reiter RJ, Herman TS. Melatonin: from basic research to cancer treatment clinics. J Clin Oncol. 2002 May 15;20(10):2575-601. doi: 10.1200/JCO.2002.11.004. PMID 12011138
- [Derived] Ramli I, Susworo S, Nuranna L, Mansyur M, Harahap AR, Soetopo S, Siregar NC, Wanandi SI. Circadian as a prognostic factor for radiation responses in patients with cervical cancer: A nested case-control study. Oncol Rep. 2022 Nov;48(5):199. doi: 10.3892/or.2022.8414. Epub 2022 Sep 23. PMID 36148886